CLINICAL TRIAL: NCT06529250
Title: A Multicenter, Randomized, Controlled Clinical Trial of Intermediate-dose HAD Regimen for CEBPA Double-mutated Acute Myeloid Leukemia
Brief Title: Intermediate-dose HAD Regimen for CEBPA Double-mutated AML
Acronym: HADCEBPA2023
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023005
Record Dates: First submitted 2024-07-17; First posted 2024-07-31 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-08

CONDITIONS: AML
Keywords: AML; CEBPA double-mutated; treatment
MeSH Terms: interventions — Homoharringtonine; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermediate-dose HAD regimen (Experimental): Patients received intermediate-dose HAD regimen. When patients reach complete remission (CR) after the induction therapy, 3 courses of the high-dose cytarabine regimen (3g/m2 q12h, 3 days) are used. Hematopoietic stem cell transplantation is recommended for patients with persistent MRD positive after treatment. When patients do not achieve CR after the induction therapy, reinduction therapy with IAC (IDA 10mg/m2 for 3 days, cytarabine 100mg/m2 for 7 days, cyclophosphamide 350mg/m2 d2, d5) regimen is used. Patients who still do not achieve CR after reinduction therapy will be removed from the group.
  Interventions: Drug: HAD
- conventional treatment (Active Comparator): Patients were treated with 3+7 induction regimen (IA or DA). When patients reach complete remission (CR) after the induction therapy, 3 courses of the high-dose cytarabine regimen (3g/m2 q12h, 3 days) are used. Hematopoietic stem cell transplantation is recommended for patients with persistent MRD positive after treatment. When patients do not achieve CR after the induction therapy, reinduction therapy with IAC (IDA 10mg/m2 for 3 days, cytarabine 100mg/m2 for 7 days, cyclophosphamide 350mg/ m2 d2, d5) regimen is used. Patients who still do not achieve CR after reinduction therapy will be removed from the group.
  Interventions: Drug: Daunorubicin+Cytarabine

INTERVENTIONS:
Drug: HAD — Induction therapy:Homoharringtonine: 2mg/㎡/d, days 1-7 Cytarabine: (Ara-c 100mg/㎡/d, day 1-4; 1g/㎡ /q12h, day 5-7), Daunorubicin: (DNR 40mg/㎡/d, day 1-3).
  Reinduction therapy:
  Idarubicin (IDA) 10mg/㎡ for d1-3 , Ara-c 100mg/㎡ d1-7 , Cyclophosphamide (CTX350mg/㎡ d2, d5) . Patients who did not achieve CR after reinduction therapy were removed from the group.
  After achieving CR, they received high-dose cytarabine (3g/m2 q12h, 3 days) regimen for consolidation for 3 courses. Hematopoietic stem cell transplantation is recommended for patients with persistent MRD positive after treatment.
  Other Names: Homoharringtonine; Cytarabine; Daunorubicin
  Arms: intermediate-dose HAD regimen
Drug: Daunorubicin+Cytarabine — Cytarabine: (Ara-c 100mg/㎡/d, day 1-7), Daunorubicin: (DNR 60mg/㎡/d, day 1-3) or idarubicin (IDA 12mg/㎡/d, day 1-3).
  Treatment did not achieve CR, and reinduction of IAC regimen was given.
  Reinduction therapy:
  Idarubicin (IDA) 10mg/㎡ ,d1-3, Ara-c 100mg/㎡ d1-7 , Cyclophosphamide (CTX350mg/㎡ d2, d5). Patients who did not achieve CR after reinduction therapy were removed from the group.
  After achieving CR, they received high-dose cytarabine (3g/m2 q12h, 3 days) regimen for consolidation for 3 courses. Hematopoietic stem cell transplantation is recommended for patients with persistent MRD positive after treatment.
  Other Names: Cytarabine; Daunorubicin
  Arms: conventional treatment

SUMMARY:
AML is highly heterogeneous in pathogenesis, and CEBPA double-mutated (CEBPAdm) AML is a common type of leukemia in China. Currently, no targeted therapies for CEBPAdm, and chemotherapy and transplantation are still the treatment options for CEBPA double-mutated AML. At present, the "3+7" treatment induction regimen of cytarabine combined with anthracyclines is still the first-line recommended regimen. In our retrospective study, the intermediate dose HAD regimen produced a 3-year RFS of 84.7% and a 3-year OS of 92.8% in CEBPAdm AML. Therefore, this project intends to confirm the efficacy of intermediate-dose HAD in the treatment of CEBPA double-mutated AML is superior to the conventional treatment regimen through the multi-center RCT study.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical trial of patients diagnosed with CEBPA double-mutated AML. Patients who meet the inclusion criteria are randomly assigned to receive the intermediate-dose HAD regimen or the conventional 3+7 induction regimen (IA or DA), respectively. When patients reach complete remission (CR) after the induction therapy, 3 courses of the high-dose cytarabine regimen (3g/m2 q12h, 3 days) are used. Hematopoietic stem cell transplantation is recommended for patients with persistent MRD positive after treatment. When patients do not achieve CR after the induction therapy, reinduction therapy with IAC (IDA 10mg/ m2 for 3 days, cytarabine 100mg/m2 for 7 days, cyclophosphamide 350mg/m2 d2, d5) regimen is used. Patients who still do not achieve CR after reinduction therapy will be removed from the group.

ELIGIBILITY:
Inclusion Criteria:

1. AML diagnosed according to WHO-2022 classification with recurrent CEBPA mutations and containing mutation in the bZIP domain.
2. Older than 14 years old and younger than 55 years old
3. Male or female.
4. The Eastern Cooperative Oncology Group Performance Status (ECOG-PS) of AML patients were 0-2 points.
5. Meet the following laboratory tests (performed within 7 days prior to treatment) 1) Total bilirubin ≤ 1.5 times of the upper limit of normal value (same age); 2) AST and ALT≤ 2.5 times of the upper limit of normal value (same age); 3) Blood creatinine < 2 times of the upper limit of normal value (same age); 4) Myocardial enzymes < 2 times of the upper limit of normal value (same age); 5) Echocardiography (ECHO) was performed to determine the ejection fraction of the heart within the normal range.

Exclusion Criteria:

1. Patients who have previously received induction chemotherapy, regardless of efficacy.
2. Simultaneously suffering from malignant tumors of other organs and requiring treatment).
3. Pregnant or lactating women. Male or female patients participating in the trial must take contraceptive measures during the trial treatment period.
4. Active heart disease, defined as one or more of the following:1) Have a history of uncontrolled or symptomatic angina pectoris;2) Myocardial infarction less than 6 months prior to enrollment in the study;3) A history of arrhythmia requiring medication treatment or severe clinical symptoms;4) Uncontrolled or symptomatic congestive heart failure (> NYHA grade 2);5) The ejection fraction is below the lower limit of the normal range.
5. Serious infectious diseases (uncured tuberculosis, pulmonary aspergillosis).
6. Those who were not considered suitable for inclusion by the researchers.

Ages: 14 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | up to 2 years after the date of the last enrolled participants
  The interval from randomization to assessment of response after the second course of chemotherapy treatment if patients failed to achieve CR after two courses of induction therapy, the date of relapse, or the date of death, whichever occurred first.

SECONDARY OUTCOMES:
Complete response rate (CR) | Six weeks after induction therapy
  The proportion that reaches CR status after two courses of induction therapy. Patients should be morphologically free of leukemia, and free of extramedullary leukemia. Absolute neutrophil counts was greater than 1.0*10^9/L, and platelet counts was greater than 100*10^9/L.
30-day mortality | Within 30 days of randomization
  Percentage of patients who died within 30 days from randomization
overall survival | up to 2 years after the date of the last enrolled participants
  The interval from the date of randomization to the date of death or the date of last follow-up for surviving patients.
Event-free survival censored at hematopoietic stem cell transplantation | up to 2 years after the date of the last enrolled participants
  The interval from randomization to assessment of response after the second course of chemotherapy treatment if patients failed to achieve CR after two courses of induction therapy, the date of relapse, or the date of death, or the date of last follow-up, or the date of hematopoietic stem cell transplantation, whichever occurred first.
Relapse free survival censored at hematopoietic stem cell transplantation | up to 2 years after the date of the last enrolled participants
  The interval from CR to the date of relapse, or the date of death, or the date of last follow-up, or the date of hematopoietic stem cell transplantation, whichever occurred first. This outcome analyze patients achieved CR in two courses induction therapy.
overall survival censored at hematopoietic stem cell transplantation | up to 2 years after the date of the last enrolled participants
  It is defined as the time from randomization to the date of death or the date of last follow-up, or the date of hematopoietic stem cell transplantation, whichever occurred first.
60-day mortality | Within 60 days of randomization
  Percentage of patients who died within 60 days from randomization
Relapse free survival(RFS) | up to 2 years after the date of the last enrolled participants
  The interval from CR to the date of relapse, or the date of death, or the date of last follow-up, whichever occurred first. This outcome analyze patients achieved CR in two courses induction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, MD, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Blood Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wei H, Wang Y, Zhou C, Lin D, Liu B, Liu K, Qiu S, Gong B, Li Y, Zhang G, Wei S, Gong X, Liu Y, Zhao X, Gu R, Mi Y, Wang J. Distinct genetic alteration profiles of acute myeloid leukemia between Caucasian and Eastern Asian population. J Hematol Oncol. 2018 Feb 10;11(1):18. doi: 10.1186/s13045-018-0566-8. PMID 29427994
- [Result] Wei H, Zhou C, Liu B, Lin D, Li Y, Wei S, Gong B, Zhang G, Liu K, Gong X, Fang Q, Liu Y, Qiu S, Gu R, Song Z, Chen J, Yang M, Zhang J, Jin J, Wang Y, Mi Y, Wang J. The prognostic factors in acute myeloid leukaemia with double-mutated CCAAT/enhancer-binding protein alpha (CEBPAdm). Br J Haematol. 2022 May;197(4):442-451. doi: 10.1111/bjh.18113. Epub 2022 Mar 10. PMID 35274287
- [Result] Wei H, Wang Y, Gale RP, Lin D, Zhou C, Liu B, Qiu S, Gu R, Li Y, Zhao X, Wei S, Gong B, Liu K, Gong X, Liu Y, Zhang G, Song Z, Wang Y, Li W, Mi Y, Wang J. Randomized Trial of Intermediate-dose Cytarabine in Induction and Consolidation Therapy in Adults with Acute Myeloid Leukemia. Clin Cancer Res. 2020 Jul 1;26(13):3154-3161. doi: 10.1158/1078-0432.CCR-19-3433. Epub 2020 Feb 6. PMID 32029439